CLINICAL TRIAL: NCT03611946
Title: Phase I Evaluation of the Safety and Immunogenicity of the Live Attenuated Zika Vaccine rZIKV/D4Δ30-713 in Flavivirus-naïve Adults
Brief Title: Safety and Immunogenicity of the Live Attenuated Zika Vaccine rZIKV/D4Δ30-713 in Flavivirus-naïve Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 318
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Zika Virus
Keywords: Zika virus; Vaccine
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Vaccine (Experimental): Single dose of rZIKV/D4Δ30-713 (10^3 PFU) via subcutaneous injection (0.5ml).
  Interventions: Biological: Single dose of rZIKV/D4Δ30-713 (10^3 PFU) via subcutaneous injection (0.5ml)
- Cohort 1 - Placebo (Placebo Comparator): Single dose of placebo via subcutaneous injection (0.5ml).
  Interventions: Biological: Single dose of placebo via subcutaneous injection (0.5ml).
- Cohort 2 - Vaccine (Experimental): Single dose of rZIKV/D4Δ30-713 (10^4 PFU) via subcutaneous injection (0.5ml).
  Interventions: Biological: Single dose of rZIKV/D4Δ30-713 (10^4 PFU) via subcutaneous injection (0.5ml)
- Cohort 2 - Placebo (Placebo Comparator): Single dose of placebo via subcutaneous injection (0.5ml).
  Interventions: Biological: Single dose of placebo via subcutaneous injection (0.5ml).

INTERVENTIONS:
Biological: Single dose of rZIKV/D4Δ30-713 (10^3 PFU) via subcutaneous injection (0.5ml) — Administered at a dose of 10^3 plaque-forming units (PFUs) by subcutaneous injection
  Arms: Cohort 1: Vaccine
Biological: Single dose of placebo via subcutaneous injection (0.5ml). — Administered by subcutaneous injection.
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo
Biological: Single dose of rZIKV/D4Δ30-713 (10^4 PFU) via subcutaneous injection (0.5ml) — Administered at a dose of using 10^4 plaque-forming units (PFUs) by subcutaneous injection.
  Arms: Cohort 2 - Vaccine

SUMMARY:
This is a phase 1 double-blind, placebo controlled trial designed to evaluate the safety, reactogenicity, and immunogenicity of a single dose of the live attenuated Zika vaccine rZIKV/D4Δ30-713 in adults with no history of previous flavivirus infection.

DETAILED DESCRIPTION:
Fifty-six healthy volunteers will be enrolled over 2 sequential cohorts:

Cohort 1: n=28, volunteers will be randomly assigned to a single dose of either vaccine (10^3 PFU, n=20) or placebo (n=8). Cohort 1 will be enrolled and evaluated first. If the vaccine is not found to induce seroconversion to ZIKV in > 80% of subjects inoculated with 10-^3 PFU of the vaccine, a second cohort of volunteers will be enrolled and will be inoculated with 10^4 PFU of vaccine (or placebo).

Cohort 2: n=28, volunteers will be randomly assigned to a single dose of either vaccine (10^4 PFU, n=20) or placebo (n=8).

All volunteers will be followed on an outpatient basis for 6 months following vaccination (13 follow up visits over 180 days). Follow up visits will include clinical assessments as well as sample collection for evaluation of viremia and seroconversion. Sample collection will include blood, urine, saliva, nasopharyngeal or midturbinate swab, vaginal secretion or semen collection on specified visit days throughout the 180 day follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, which is approximately 26 weeks.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females only: Female subjects of childbearing potential, with the exception noted below, should be willing to use effective contraception and have no plans to undergo IVF (in vitro fertilization) during participation in the trial. Reliable methods of contraception include hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, and intrauterine device. Women must have been on an effective method of birth control for at least 30 days prior to enrollment. All female subjects will be considered as having childbearing potential, except for women who exclusively have sex with women, those who have had a hysterectomy, tubal ligation, or tubal coil (at least 3 months prior to vaccination), or are considered to be post-menopausal, as documented by at least 1 year since last menstrual period with a follicle-stimulating hormone (FSH) level in the menopausal range or at least 24 consecutive months of amenorrhea. Transgender men who have internal female organs and have sex with men will be considered of childbearing potential and should be willing to use effective contraception during the trial. Exception: Females who have sex with females (exclusively) and have no intention of conceiving a child during the study and women whose partners have had a vasectomy will not be required to use contraception, however they will be required to use female condoms and/or dental dams for at least 1 month following vaccination. For women whose sexual partner has had a vasectomy, the vasectomy must have been performed 30 days or more prior to enrollment.
* Males only: Males of reproductive potential should be willing to use barrier contraception for the first 3 months following vaccination* and agree to not donate sperm for the duration of the study.

  * Based on CDC guidance for men returning from ZIKV-endemic areas

Exclusion Criteria:

* Females only: Currently pregnant, as determined by positive β-human choriogonadotropin (HCG) test, or breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the requirements of the study protocol.
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol.
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, as indicated by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, as indicated by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, as indicated by hepatitis B surface antigen (HBsAg) screening.
* Any known immunodeficiency syndrome.
* History of Guillain-Barrè syndrome.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of immunosuppressive corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following inoculation. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg of a prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within 14 days prior to inoculation, or anticipated receipt of any vaccine during the 28 days following inoculation with the exception of COVID-19 vaccines either licensed or under EUA which can be given at any time, however all effort will be made to avoid giving COVID-19 vaccines within the above windows.
* Asplenia.
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following inoculation.
* History or serologic evidence of previous ZIKV or other flavivirus infection (e.g., dengue, yellow fever virus, St. Louis Encephalitis virus, or West Nile virus).
* Previous receipt of a flavivirus vaccine (licensed or experimental).
* Receipt or anticipated receipt of any investigational agent in the 28 days before or after inoculation with the exception of COVID-19 vaccines, either licensed or authorized under EUA.
* Refusal to allow specimen storage for future research.
* Is in isolation or quarantine for SARS-CoV-2 infection or exposure and cannot complete screening or enrollment for this reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health; Kristen Pierce, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland
  - University of Vermont Medical Center (UVMMC), Clinical Research Center, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Vaccine: Single dose of rZIKV/D4Δ30-713 (10^3 PFU) administered via subcutaneous injection (0.5ml).
- Cohort 1 - Placebo; Cohort 2 - Placebo: Single dose of placebo administered via subcutaneous injection (0.5ml).
- Cohort 2 - Vaccine: Single dose of rZIKV/D4Δ30-713 (10^4 PFU) administered via subcutaneous injection (0.5ml)
Period: Overall Study
Arm/Group | Cohort 1 - Vaccine | Cohort 1 - Placebo | Cohort 2 - Vaccine | Cohort 2 - Placebo
Started | 20 | 8 | 20 | 8
Completed | 20 | 8 | 19 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - Vaccine: rZIKV/D4Δ30-713 (10^3 PFU) via subcutaneous injection (0.5ml).
- Cohort 1 - Placebo; Cohort 2 - Placebo: Administered via subcutaneous injection (0.5ml).
- Cohort 2 - Vaccine: rZIKV/D4Δ30-713 (10^4 PFU) via subcutaneous injection (0.5ml)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Vaccine | Cohort 1 - Placebo | Cohort 2 - Vaccine | Cohort 2 - Placebo | Total
Number analyzed (Participants) | 20 | 8 | 20 | 8 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 8 | 20 | 8 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 17 | 6 | 37
  Male | 11 | 3 | 3 | 2 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 3 | 2 | 11
  White | 14 | 5 | 14 | 6 | 39
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
PRNT (50) ZIKV <= 10 [Count of Participants; unit: Participants] — PRNT (50) is defined as the highest dilution of antibody that reduces the number of foci or plaques by 50% compared to the plaque titer of the virus [ZIKV] alone. [Indicator of prior exposure to ZIKV].
  Participants | 20 | 8 | 20 | 8 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and General Adverse Events (AEs)
Description: Evaluated using the Adverse Event Grading Table in the study protocol.
Time Frame: Solicited AE's assessed every visit through Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - Vaccine: rZIKV/D4Δ30-713 (10^3 PFU) administered via subcutaneous injection (0.5ml)
- Cohort 1 Placebo; Cohort 2 Placebo: Placebo administered via subcutaneous injection (0.5ml)
- Cohort 2 - Vaccine: rZIKV/D4Δ30-713 (10^4 PFU) administered via subcutaneous injection (0.5ml)
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 8 | 20 | 8
Participants
  headache | 10 | 5 | 8 | 5
  fatigue | 5 | 2 | 4 | 2
  nausea | 4 | 2 | 2 | 2
  myalgia | 4 | 2 | 3 | 2
  arthralgia | 2 | 1 | 2 | 0
  retro-orbital pain (ROP) | 1 | 1 | 0 | 2
  photophobia | 1 | 0 | 1 | 0
  injection site erythema | 1 | 0 | 1 | 0
  muscle weakness | 1 | 0 | 0 | 0
  fever | 0 | 0 | 1 | 0
  Zika-like rash | 0 | 0 | 0 | 0
  elevated ALT | 0 | 0 | 0 | 0
  Neutropenia | 0 | 0 | 0 | 0
  Thrombocytopenia | 0 | 0 | 0 | 0
  Injection Site Pain | 0 | 0 | 0 | 0
  Injection Site Tenderness | 0 | 0 | 0 | 0
  Injection Site Induration | 0 | 0 | 0 | 0
  Injection Site Pruritus | 0 | 0 | 0 | 0
  prolonged PT | 0 | 0 | 0 | 0
  prolonged PTT | 0 | 0 | 0 | 0

2. Primary Outcome: To Determine the Immunogenicity of a Single Dose of rZIKV/D4Δ30-713
Description: Determination of the serum plaque reduction neutralization titer 50% (PRNT50) to ZIKV for each subject at Study Day 28 post-inoculation. Seroconversion will be defined as achieving a PRNT50 ≥ 1:10 at any time-point through Study Day 28. The peak PRNT50 to ZIKV through Study Day 28 will be calculated for each subject included in the per-protocol an intent-to-treat analysis and the geometric mean peak titer for vaccinated subjects will be calculated.
Time Frame: Measured through Day 28
Population: Note "titer" is not available under "measure type" option. Therefore we went with the best-fitting answer of "number".
Measure: Geometric Mean (Full Range); unit: PRNT(50) Titer
Arm/Group | Cohort 1 - Vaccine | Cohort 2 - Vaccine
Number analyzed (Participants) | 20 | 19
PRNT(50) Titer | 56.1 [12.3 to 59.2] | 126.1 [49.8 to 320]

3. Secondary Outcome: Viremia Induced by Vaccine (Number of Participants With Detectable Virus at Any Time Point)
Description: Assess the frequency, quantity, and duration of viremia (virus in the blood) induced by a single dose of the rZIKV/D4Δ30-713 vaccine. The mean peak viremia, mean day of onset of viremia, and mean duration of viremia will be calculated. Viremia will be detected by culture (infectious virus) and by RT-PCR.
Time Frame: Measured through Day 90
Population: Analysis that is applicable only to post-vaccine (not placebo) subjects.
Measure: Number; unit: #participants w/ vaccine-induced viremia
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 0 | 19 | 0
#participants w/ vaccine-induced viremia | 0 |  | 0 |

4. Secondary Outcome: Number of Vaccinees Infected With rZIKV/D4Δ30-713
Description: Determine the number of vaccinees infected with rZIKV/D4Δ30-713. Infection is defined as recovery of infectious vaccine virus from the blood, serum or urine of a subject and/or by seroconversion to ZIKV. Seroconversion will be defined as achieving a PRNT50 ≥ 1:10 by Study Day 90 post-vaccination.
Time Frame: Measured through Day 180
Population: Analysis that is applicable only to post-vaccine (not placebo) subjects.
Measure: Number; unit: #participants who seroconverted
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 0 | 19 | 0
#participants who seroconverted | 9 |  | 7 |

5. Secondary Outcome: Immunogenicity of rZIKV/D4Δ30-713 in Flavivirus-naïve Subjects
Description: Evaluate the immunogenicity of rZIKV/D4Δ30-713 in flavivirus-naïve subjects as assessed by the PRNT50 to ZIKV, for each subject at Study Day 28, 56, and 90 post-administration of LA Zika vaccine. Expressed as geometric mean peak titer, reciprocal (median). Geometric mean titer was calculated at each time point for only those subjects with a titer of >= 10, reciprocal. Seroconversion was defined as a PRNT(50) of >= 10, reciprocal.
Time Frame: Measured through Day 180
Population: Analysis that is applicable only to post-vaccine (not placebo) subjects.
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 0 | 19 | 0
titer | 56.1 [12.3 to 59.2] |  | 126.1 [15.2 to 320] |

6. Secondary Outcome: Durability of Antibody Response
Description: Determine the durability of antibody response 26 weeks after vaccination. Neutralizing antibody titers to ZIKV were measured at 0, 28, 56, 90, 150, and 180 days following vaccination, with the peak neutralizing antibody titer determined as the peak titer in the 90 days following vaccination for either dose cohort.
Time Frame: 26 Weeks post vaccination
Population: Analysis that is applicable only to post-vaccine (not placebo) subjects.
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 0 | 19 | 0
titer | 56.1 [12.3 to 59.2] |  | 126.1 [15.2 to 320] |

7. Secondary Outcome: Quantity and Duration of ZIKV Presence
Description: Determine the quantity and duration of ZIKV presence as determined by:
  * The peak virus titer in the blood and the duration of viremia induced by the LA Zika vaccine as determined by RT-PCR and virus culture
  * The quantity and duration of possible Zika vaccine shedding in urine determined by RT-PCR and virus culture
  * The quantity and duration of possible Zika vaccine shedding in vaginal secretions determined by RT-PCR and virus culture
  * The quantity and duration of possible Zika vaccine shedding in semen determined by RT-PCR and virus culture
Time Frame: 90 days post vaccination
Population: Number of participants with recovered ZIKV from any bodily fluid (serum, urine, semen, and cervico-vaginal secretions) at any time point post-vaccination, as assessed by PCR and culture.
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1 - Vaccine | Cohort 1 Placebo | Cohort 2 - Vaccine | Cohort 2 Placebo
Number analyzed (Participants) | 20 | 8 | 19 | 8
Number of participants
  Recovered vaccine virus from serum at any time point post-vaccination as assessed by PCR and culture | 0 | 0 | 0 | 0
  Recovered vaccine virus from urine at any time point post-vaccination as assessed by PCR and culture | 0 | 0 | 0 | 0
  Recovered vaccine virus from semen at any time point post-vaccination as assessed by PCR and culture: number analyzed (Participants) | 11 | 3 | 3 | 2
  Recovered vaccine virus from semen at any time point post-vaccination as assessed by PCR and culture | 0 | 0 | 0 | 0
  Recovered vaccine virus from CVS at any time point post-vaccination as assessed by PCR and culture: number analyzed (Participants) | 9 | 5 | 16 | 6
  Recovered vaccine virus from CVS at any time point post-vaccination as assessed by PCR and culture | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs will be evaluated for severity, action taken, seriousness, outcome, and relationship to the investigational vaccine as described in Section 8.2 in this protocol. AEs will be collected through the 28- day period following inoculation, and any test agent-related AEs (adverse reactions) identified in the 28-day post-inoculation period will be followed until resolution.
Groups:
- Cohort 1 - Placebo; Cohort 2 - Placebo: Placebo administered via subcutaneous injection (0.5ml)
Arm/Group | Cohort 1 - Vaccine | Cohort 1 - Placebo | Cohort 2 - Vaccine | Cohort 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/8 | 0/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 1/20 | 0/8
Other Adverse Events (participants affected / at risk) | 14/20 | 6/8 | 11/20 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Vaccine (N=20) | Cohort 1 - Placebo (N=8) | Cohort 2 - Vaccine (N=20) | Cohort 2 - Placebo (N=8)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA — Stage 1 breast female cancer. Event preventing daily activity and requiring medical intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Vaccine (N=20) | Cohort 1 - Placebo (N=8) | Cohort 2 - Vaccine (N=20) | Cohort 2 - Placebo (N=8)
Headache (General disorders) | 10 | 5 | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Retroorbital pain (Eye disorders) | 1 | 1 | 0 | 2
Fatigue (General disorders) | 5 | 2 | 4 | 2
Nausea (Gastrointestinal disorders) | 4 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03611946/Prot_SAP_001.pdf